CLINICAL TRIAL: NCT01837953
Title: Stepped Care for Binge Eating Disorder: Predicting Response to Minimal Intervention in a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120689-01H
Record Dates: First submitted 2013-01-28; First posted 2013-04-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unguided Self-Help, No Further Treatment for 16 Weeks (Other): All participants will first receive 10 weeks of unguided self-help (USH), followed by no further treatment for 16 weeks. Participants will be offered a follow up referral to the eating disorders program at The Ottawa Hospital after the 16 week no-treatment period.
  Interventions: Behavioral: Unguided Self-Help
- Unguided Self-Help, GPIP (Experimental): All participants will first receive 10 weeks of unguided self-help (USH). For those participants randomized to the USH + Group Psychodynamic Interpersonal Psychotherapy condition, this second step will consist of 16 weekly 90 minute sessions of Group Psychodynamic Interpersonal Psychotherapy.
  Interventions: Behavioral: Group Psychodynamic Interpersonal Psychotherapy; Behavioral: Unguided Self-Help

INTERVENTIONS:
Behavioral: Group Psychodynamic Interpersonal Psychotherapy — For those participants randomized to the USH + Group Psychodynamic Interpersonal Psychotherapy (GPIP) condition, this intervention will consist of 16 weekly 90 minute sessions of GPIP. GPIP was developed and empirically tested in a randomized controlled trial (RCT) at our Centre. GPIP will be preceded by an individual pre-group preparation session conducted by a psychologist trained in GPIP to orient the patient to the therapy. Patients are given a rationale for the treatment. Examples of the patient's cyclical relational patterns (CRPs) that may underlie their symptoms are discussed and the patient will be encouraged to work on these in the groups. Therapists will be given a written summary of each patient's CRP.
  Arms: Unguided Self-Help, GPIP
Behavioral: Unguided Self-Help — All participants will first receive 10 weeks of Unguided Self-help. The USH will be based on Dr. Christopher Fairburn's CBT-oriented and evidence based self-help treatment plan for binge eating explained in his book, Overcoming Binge Eating. The USH program follows six steps: (1) Getting Started: Self-monitoring, weekly weighing; (2) Regular Eating: Establishing a pattern of regular eating; (3) Alternatives to Binge Eating: Substituting alternative activities; (4) Problem Solving and Taking Stock: Practicing problem solving and reviewing progress; (5) Dieting and Related Forms of Avoidance: Tackling the three forms of dieting and other forms of avoidance eating; and (6) What Next? Preventing relapse and dealing with other problems.

SUMMARY:
Binge Eating Disorder (BED) affects as many as 3% of women and men in Ontario, 8% of obese individuals, and 30% to 50% of those participating in weight loss programs. BED, the most common eating disorder, is characterized by over-eating with loss of control (i.e., binge eating), but with no purging (e.g., vomiting).Our previous research indicates that the total health care costs for women with BED is 36% higher than the Canadian average for women of a similar age, and that health care costs significantly decreased following intensive treatment at our Centre. The main goal of our study is to inform the development of a stepped care approach to the treatment of BED. Stepped care involves providing easily accessible low intensity treatment first, and then providing more expensive intensive treatment second, if necessary. The second goal is to assess if a second more intensive step of treatment provides added value. Although stepped care for BED is suggested by a number of clinicians and researchers, no study adequately tests predictors of who might benefit from minimal treatment alone and who would require the more intensive second step. The results of this study will guide decision making regarding who benefits from stepped care, and will help to increase the accessibility, availability, and cost effectiveness of psychological treatments for BED.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they:

  1. are comfortable speaking or reading English;
  2. do not have a history of an eating disorder other than BED, or a history of significant purging behaviour;
  3. do not have a concurrent DSM-IV diagnosis of bipolar disorder, psychosis, drug or alcohol dependence;
  4. are not currently or planning to be enrolled in a weight-loss program within the next year;
  5. are women who are not pregnant or planning to be pregnant within the next year; and
  6. are not currently or planning to be enrolled in other psychotherapies within the next year

Exclusion Criteria:

* Participants will be excluded if they:

  1. are not comfortable speaking or reading English;
  2. have a history of an eating disorder other than BED, or a history of significant purging behaviour;
  3. have a concurrent DSM-IV diagnosis of bipolar disorder, psychosis, drug or alcohol dependence;
  4. are currently or plan to be enrolled in a weight-loss program within the next year;
  5. are women who are pregnant or planning to be pregnant within the next year; and
  6. are currently or plan to be enrolled in other psychotherapies within the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Binge Eating Episodes in the Past 28 Days. | Up to one and a half years
  Binge eating is assessed in a structured interview using a calendar recall method (Wilfley et al., 1993).

SECONDARY OUTCOMES:
Body Mass Index (BMI). | Up to one and a half years
  This outcome variable will be calculated by dividing weight (kg) by height (m2).
Center for Epidemiologic Studies Depression Scale (CES-D) | Up to one and a half years
  The CES-D is a brief self-report measure of depressive symptoms.
Experiences in Close Relationships Scale (ECR) | Up to one and a half years
  The ECR, a predictor of USH outcome, is a 36-item measure comprising two 18-item scales (Avoidance and Anxiety). Items are scored on a 7-point Likert scale, ranging from 1 = Disagree Strongly to 7 = Agree Strongly.
Inventory of Interpersonal Problems (IIP-64) | Up to one and a half years
  The IIP-64 assesses interpersonal problems; higher scores indicate greater problems. The IIP is a 64-item scale with a 5-point Likert-type response format.
Patient Health Questionnaire 9 (PHQ-9). | Up to one and a half years
  The PHQ-9 is a 9-item self-report measure. The PHQ-9 is used in assessing the severity of depressive symptomology and can act as a diagnostic tool (Kroenke et al., 2001).
Rapid Response to Treatment: Self-Monitoring | From the date of the start of unguided self-help to the end of self-help (Up to 10 weeks)
  Self monitoring of binge eating is an indicator of rapid response to USH, which is a predictor of USH outcome. Daily record sheets will be used to assess objective binge eating episodes on an on-going basis throughout the course of USH. In each daily record, participants record whether they had any overeating behaviors (including objective binge episodes) and how many. The daily record forms provide a definition of objective binge episodes based on the EDE definition. These definitions will be reviewed with participants at the start of USH.
Rosenberg Self Esteem Scale (RSES) | Up to one and a half years
  The RSES, a predictor of USH outcome and an outcome variable, will be used to measure self esteem. The RSES is a ten-item self-report scale using a four-point response format. Scores are summed to produce a total score ranging from 0 to 30, with higher scores representing higher self esteem.
Eating Disorder Diagnostic Scale (EDDS) | From the start of Group Psychodynamic Interpersonal Psychotherapy (GPIP) to the end of GPIP (Up to 16 weeks)
  This is a self report measure of eating disorder symptoms including binge eating
Experiences in Close Relationships Scale Short Form (ECR-S). | From the start of Group Psychodynamic Interpersonal Psychotherapy (GPIP) to the end of GPIP (Up to 16 weeks)
  The ECR-S, a predictor of USH outcome, is a 12-item measure comprising two 6-item scales (Avoidance and Anxiety). Items are scored on a 7-point Likert scale, ranging from 1 = Disagree Strongly to 7 = Agree Strongly. The ECR-S was derived from the full ECR scale which was derived from existing self-report adult romantic attachment measures.
Therapeutic Factors Inventory (TFI) | From the start of Group Psychodynamic Interpersonal Psychotherapy (GPIP) to the end of GPIP (Up to 16 weeks)
  The full 99-item TFI will not be used in its entirety but rather the 9-item subscale of cohesiveness will only be used to measure levels of group cohesion throughout GPIP. It is a 7-point Likert-type scale with responses ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
Outcome Rating Scale (ORS) | From the start of Group Psychodynamic Interpersonal Psychotherapy (GPIP) to the end of GPIP (Up to 16 weeks)
  The ORS was originally developed as a shorter form of the Outcome Questionnaire 45.2 (Miller et al., 2003). The ORS is a 4-item self-report scale that will be used as a treatment outcome measure of GPIP.
Working Alliance Inventory Short (WAI-S). | From the start of Group Psychodynamic Interpersonal Psychotherapy (GPIP) to the end of GPIP (Up to16 weeks)
  The WAI is a 12-item self-report measure of alliance to therapist and in this case the GPIP therapist.
Eating Disorder Examination - Questionnaire (EDE-Q) | Up to one and a half years
  The EDE-Q, an outcome scale, is a 28-item self-report measure modeled on the EDE interview (Fairburn & Cooper, 1993). The EDE-Q Restraint scale measures dietary restraint, Eating Concern scale measures concern about eating, Shape Concern scale measures preoccupation with one's body shape, and Weight Concern scale measures preoccupation with one's body weight (Fairburn & Beglin, 1994)). The EDE-Q also provides a single overall score of eating disorder psychopathology based on the scales.
Depression Anxiety and Stress Scales 21(DASS-21) | Up to one and a half years
  The DASS-21 is a self-report measure of stress, anxiety, and depression.

CONTACTS AND LOCATIONS:
Overall Officials: George A Tasca, Ph.D,C.Psych, Principal Investigator — University of Ottawa, Ottawa Hospital: General Campus
Locations (1):
- Regional Centre for the Treatment of Eating Disorders, Ottawa, Ontario, Canada